CLINICAL TRIAL: NCT03259035
Title: NEO: Neoadjuvant Chemotherapy, Excision and Observation for Early Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO28
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Intervention Model Description: This is a two staged, single arm phase II trial of chemotherapy (FOLFOX or CAPOX) followed by tumour excision in patients with early stage rectal cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- chemotherapy (FOLFOX or CAPOX) followed by tumour excision (Experimental)
  Interventions: Drug: Folfox Protocol; Drug: Capox

INTERVENTIONS:
Drug: Folfox Protocol — 6 cycles of q2weekly FOLFOX, or
Drug: Capox — 4 cycles of q3weekly CAPOX

SUMMARY:
The purpose of this study is to find out the effects of chemotherapy followed by less invasive surgery on patients and their early rectal cancer. The approach of this trial will be considered a success if at least 65% of participants are able to keep the rectum.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive well-moderately differentiated rectal adenocarcinoma diagnosed within 90 days prior to enrollment.
* Tumour stage cT1-T3abN0 based on pelvic MRI

  * cT1N0- tumour invasion into submucosa, no radiographic evidence of mesorectal nodal metastasis, tumour deposits or vascular invasion.
  * cT2N0 - tumour invasion into muscularis propria, no radiographic evidence of mesorectal nodal metastasis, tumour deposits or vascular invasion.
  * cT3a,bN0- tumour invasion through the muscularis propria no more than 5 mm into the subserosa/perirectal tissue and clear of the circumferential radial margin (CRM). Absence of radiographic evidence of mesorectal nodal metastasis, tumour deposits or lymphovascular invasion.

Note: If the tumour is not visualized in the MRI but there is histological confirmation of rectal adenocarcinoma the patient is eligible.

* cN0 stage based on pelvic MRI. Any nodes ≥ 10 mm in longest dimension are considered malignant, regardless of nodal morphology. For pelvic nodes < 10 mm in longest dimension, if nodes are seen and are deemed to be morphologically benign in the opinion of the radiologist and surgeon, the patient is eligible. Patients with visible pelvic sidewall nodes are excluded
* M0 stage based on no evidence of metastatic disease by CT imaging.
* Mid to low-lying tumour eligible for local tumour excision in the opinion of the treating surgeon.
* Age of at least 18 years.
* Medically fit to undergo radical surgery as per treating surgeon's discretion
* No contraindications to protocol chemotherapy.
* Adequate normal organ and marrow function as defined below (must be done within 30 days prior to enrolment):

  * ANC ≥ 1.5 x 109/L
  * platelet count ≥100 x 109/L
  * bilirubin < 1.5 ULN, excluding Gilbert's syndrome
  * Calculated creatinine clearance of ≥ 50 ml/min.
  * Clearance to be calculated using Cockcroft formula: Males: 1.23 x (140 - age) x weight (kg) - serum creatinine (μmol/l) ; Females: 1.05 x (140 - age) x weight (kg) - serum creatinine (μmol/l)
* The patient must have an ECOG performance status of 0, 1.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life and health utility questionnaires.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Must be accessible for treatment and follow up. Patients registered on this trial must be treated with chemotherapy and followed at the enrolling centre.
* Protocol treatment is to begin within 5 working days of patient enrollment.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method during and for 6 months after completion of chemotherapy.

Exclusion Criteria:

* Patient has pathologic high risk factors on either the initial biopsy specimen report or follow-up biopsy (if done): high histologic grade, mucinous histology, lymphatic or vascular invasion.
* History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Synchronous cancer.
* Prior treatment for rectal cancer.
* Previous pelvic radiation for any reason.
* Patients with known dihydropyrimidine dehydrogenase deficiency
* Treatment with other investigational drugs or anti-cancer therapy within 28 days prior to enrolment.
* Clinically significant (i.e. active) cardiovascular disease for example cerebro vascular accidents (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, New York Heart Association (NYHA) grade II or higher, congestive heart failure, serious cardiac arrhythmia requiring medication.
* Any contra-indications to undergo MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, Study Chair — Virginia Mason Medical Centre, WA USA; Carl Brown, Study Chair — St. Paul's Hospital, Vancouver BC
Locations (11):
- United States (3):
  - UC Irvine Medical Center, Orange, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (8):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Research Institute of the McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kennecke HF, O'Callaghan CJ, Loree JM, Moloo H, Auer R, Jonker DJ, Raval M, Musselman R, Ma G, Caycedo-Marulanda A, Simianu VV, Patel S, Pitre LD, Helewa R, Gordon VL, Neumann K, Nimeiri H, Sherry M, Tu D, Brown CJ. Neoadjuvant Chemotherapy, Excision, and Observation for Early Rectal Cancer: The Phase II NEO Trial (CCTG CO.28) Primary End Point Results. J Clin Oncol. 2023 Jan 10;41(2):233-242. doi: 10.1200/JCO.22.00184. Epub 2022 Aug 18. PMID 35981270

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision: FOLFOX infusion on a 14 day cycle (IV oxaliplatin 85 mg/m2 and leucovorin 400 mg/m2 over 2 hours on day 1 and bolus fluorouracil 400 mg/m2 over 5 - 15 minutes and continuous infusion of fluorouracil 2400 mg/m2 over 46 to 48 hours on days 1-2) for a total of 6 cycles or CAPOX on a 21 day cycle (IV oxaliplatin 130 mg/m2 over 2 hours on day 1 and 1000 mg/m2 capecitabine orally twice daily for 14 days from day 1) for a total of 4 cycles.
Period: Stage 1: Chemotherapy
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Started | 58
Completed | 58
Not Completed | 0
Period: Stage 2: Tumor Excision
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in this study.
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 66.5 [31.0 to 83.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 54
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Organ Preservation
Description: Defined as the percentage of patients with tumour downstaging to ypT0/T1good N0 and who avoid radical surgery.
Time Frame: 3 years
Population: All participants who had chemotherapy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Number analyzed (Participants) | 58
percentage of participants | 57 [45 to 68]

2. Secondary Outcome: Percentage of Locoregional Relapses at 3 Years
Description: Locoregional relapse is defined as reappearance of a tumour within the rectum or pelvis. The percentage of loco-reginal relapse at 3 years was estimated by Kaplan-Meier method for the survival function of the loco-regional relapse free survival, defined as the time from enrollment to the first date of definitive evidence (clinical, radiological or pathological) of locoregional relapses with patients who developed distant relapse only, died, loss to follow up, or were alive at clinical cut-off censored at respectively at last date of distant relapses, date of death, date of lost to follow-up, or last disease assessment date.
Time Frame: 3 years
Population: All patients enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Number analyzed (Participants) | 58
percentage of participants | 7.1 [2.7 to 17.7]

3. Secondary Outcome: Percentage of Distant Relapse at 3 Years
Description: Distant relapse is defined as appearance of rectal cancer disease at sites remote from the rectum. The percentage of distant relapse at 3 years was estimated also by Kaplan-Meier method for the survival function of the distant free survival, defined as the time from enrollment to the first date of definitive evidence (clinical, radiological or pathological) of distant relapses with patients who died, loss to follow up, or were alive at clinical cut-off censored at respectively: date of death, date of lost to follow-up, and last disease assessment date.
Time Frame: 3 years
Population: All participants enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Number analyzed (Participants) | 58
percentage of participants | 5.3 [1.7 to 15.4]

4. Secondary Outcome: Percentage of Disease Free at 3 Years
Description: Percentage of disease free at 3 years was estimated by Kaplan-Meier method for the survival function of Disease-Free Survival (DFS), which is defined as the interval from date of enrollment to the first date of the events defined below:
  * Locoregional relapse
  * Distant relapse
  * Non-protocol radiotherapy, chemotherapy, or biologic therapy without documentation of the site of failure
  * Death due to any other reason. Patients who were alive without locoregional or distant relapse or receiving non-protocol radiotherapy, chemotherapy, or biologic therapy without documentation of the site of failure at the clinical data cutoff date were censored at their last disease assessment date.
    3 year disease free survival was estimated by Kaplan-Meier method.
Time Frame: 3 years
Population: All participants enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Number analyzed (Participants) | 58
percentage of participants | 84.3 [72.0 to 91.5]

5. Secondary Outcome: Rate of Intraoperative Complications
Description: Percentage of patients with at least one intraoperative injury
Time Frame: 1 day
Population: Patients who had BOTH chemotherapy and tumor excision with transanal endoscopic microsurgery (TEM) or transanal minimally invasive surgery (TAMIS)
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
Number analyzed (Participants) | 53
percentage of participants | 1.89

ADVERSE EVENTS:
Time Frame: During chemotherapy treatment (maximum 24 weeks)
Arm/Group | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision
All-Cause Mortality (participants affected / at risk) | 2/58
Serious Adverse Events (participants affected / at risk) | 1/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision (N=58)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (FOLFOX or CAPOX) Followed by Tumour Excision (N=58)
Watering eyes (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 11
Bloating (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 24
Diarrhea (Gastrointestinal disorders) | 32
Dyspepsia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9
Mucositis oral (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 42
Other gastrointestinal disorders (Gastrointestinal disorders) | 5
Rectal hemorrhage (Gastrointestinal disorders) | 19
Rectal pain (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 13
Facial pain (General disorders) | 6
Fatigue (General disorders) | 45
Fever (General disorders) | 5
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 5
Skin infection (Infections and infestations) | 3
Weight loss (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 24
Dehydration (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle cramp (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 4
Dysesthesia (Nervous system disorders) | 16
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 10
Paresthesia (Nervous system disorders) | 20
Peripheral sensory neuropathy (Nervous system disorders) | 37
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Urinary frequency (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 8
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Other skin and subcutaneous tissue disorders (Respiratory, thoracic and mediastinal disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT03259035/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT03259035/SAP_001.pdf